CLINICAL TRIAL: NCT02758392
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose, Interventional Study of JNJ-61178104 in Healthy Subjects
Brief Title: A Study to Evaluate Safety and Tolerability of JNJ-61178104 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108162; 61178104NAP1001 (Other: Janssen Research & Development, LLC); 2015-004253-40 (EudraCT Number)
Record Dates: First submitted 2016-04-14; First posted 2016-05-02 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
Keywords: Healthy; JNJ-61178104; Placebo; Safety

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Dose 1: JNJ-61178104 OR Placebo IV (Experimental): Participants will receive either JNJ-61178104 0.1 milligram/kilogram (mg/kg) or Placebo Intravenously (IV) on Day 1.
  Interventions: Drug: JNJ-61178104 Intravenous; Drug: Placebo
- Dose 2: JNJ-61178104 OR Placebo IV (Experimental): Participants will receive either JNJ-61178104 0.3 mg/kg or Placebo IV on Day 1.
  Interventions: Drug: JNJ-61178104 Intravenous; Drug: Placebo
- Dose 3: JNJ-61178104 OR Placebo IV (Experimental): Participants will receive either JNJ-61178104 1 mg/kg or Placebo IV on Day 1.
  Interventions: Drug: JNJ-61178104 Intravenous; Drug: Placebo
- Dose 4: JNJ-61178104 OR Placebo IV (Experimental): Participants will receive either JNJ-61178104 3 mg/kg or Placebo IV on Day 1.
  Interventions: Drug: JNJ-61178104 Intravenous; Drug: Placebo
- Dose 5: JNJ-61178104 OR Placebo IV (Experimental): Participants will receive either JNJ-61178104 10 mg/kg or Placebo IV on Day 1.
  Interventions: Drug: JNJ-61178104 Intravenous; Drug: Placebo
- Dose 6: JNJ-61178104 OR Placebo SC (Experimental): Participants will receive either JNJ-61178104 1 mg/kg or Placebo Subcutaneously (SC) on Day 1.
  Interventions: Drug: JNJ-61178104 Subcutaneous; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-61178104 Intravenous — Participants will receive JNJ-61178104 Intravenously on Day 1.
  Arms: Dose 1: JNJ-61178104 OR Placebo IV; Dose 2: JNJ-61178104 OR Placebo IV; Dose 3: JNJ-61178104 OR Placebo IV; Dose 4: JNJ-61178104 OR Placebo IV; Dose 5: JNJ-61178104 OR Placebo IV
Drug: JNJ-61178104 Subcutaneous — Participants will receive JNJ-61178104 Subcutaneously on Day 1.
  Arms: Dose 6: JNJ-61178104 OR Placebo SC
Drug: Placebo — Participants will receive placebo on Day 1.

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics (PK) and immunogenicity of JNJ-61178104 following a single ascending Intravenous (IV) dose administration and a single Subcutaneous (SC) dose administration in healthy participants.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, single ascending dose, single site, interventional study. There will be 5 single ascending dose (SAD) IV cohorts and 1 SC cohort. Nine participants will be enrolled into each of 5 IV cohorts and 1 SC cohort and participants will be randomized at a ratio of 2:1 to receive JNJ-61178104 or placebo. The total duration of participants participation will be approximately 21 weeks including a Screening Visit up to 4 weeks prior to study drug administration. Participants will have an inpatient period consisting of 6 days/5 nights and will return to the study-site at Weeks 2, 3, 4, 5, 7, 9, 13, and 17. Participants will be evaluated for safety throughout the study.

ELIGIBILITY:
Inclusion Criteria

* Participant must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study
* Participant must have a body weight in the range of 50 Kilogram (kg) to 100 kg, inclusive, and have a body mass index of 19 Kilogram per meter square (kg/m^2) to 30 kg/m2, inclusive
* Participant must be healthy on the basis of clinical laboratory tests performed at Screening and Day-1. If the results of the serum chemistry panel including liver enzymes, hematology panel, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's medical record with documented review confirmation by the investigator
* Before randomization, a woman must not be of childbearing potential: a) Postmenopausal {greater than (>) 45 years of age with amenorrhea for at least 12 months or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone (FSH) level >40 International Units Per Litre (IU/L) at Screening}; or b) Permanently sterilized (example, bilateral tubal occlusion, hysterectomy, bilateral salpingectomy, oophorectomy); or c) Otherwise be incapable of pregnancy
* Be considered eligible according to the following tuberculosis (TB) Screening criteria: a) Have no history of latent or active TB prior to Screening; b) Have no signs or symptoms suggestive of active TB upon medical history and/or physical examination; c) Have had no recent close contact with a person with active TB; d) Have a negative T-Spot TB test result at Screening

Exclusion Criteria:

* Participant currently has or has a history of any clinically significant medical illness or medical disorders the investigator considers should exclude the participant, including (but not limited to), neuromuscular, hematological disease, immune deficiency state, cardiac, vascular, metabolic, endocrine, rheumatologic, respiratory disease, hepatic or gastrointestinal disease, neurological or psychiatric disease, ophthalmological disorders, neoplastic disease, renal or urinary tract diseases, or dermatological disease
* Participant has a QT corrected according to Fridericia's formula (QTcF) interval >450 msec, has a complete left or right bundle branch block, or has a history or current evidence of additional risk factors for torsades de pointes (example, heart failure, hypokalemia, family history of Long QT Syndrome) at Screening and at Day -1
* Participant has had major surgery, (example, requiring general anesthesia) within 4 months before Screening, or will not have fully recovered from surgery, or has surgery planned during the time the participant is expected to participate in the study or within 17 weeks after the last dose of study drug administration
* Participant plans to undergo non-major elective surgery within 4 weeks prior to study drug administration through the end of the study
* Participant has a known or suspected intolerance or hypersensitivity to any biologic medication or known allergies or clinically significant reactions to murine, chimeric, or human proteins, monoclonal antibodies or antibody fragments, or to any components of the formulation of JNJ-61178104 and its excipients used in this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2016-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events Following Study Drug Administration as a Measure of Safety and Tolerability | Day 113

SECONDARY OUTCOMES:
Serum Concentration of JNJ-61178104 | Up to Day 113
JNJ-61178104 Antibodies Concentration | Up to Day 113
Cytokine Concentrations | Predose, Up to Day 113
Maximum Observed Serum Concentration (Cmax) Following Intravenous (IV) and Subcutaneous (SC) JNJ-61178104 Administration | Up to Day 113
Area Under the Serum Concentration-Time Curve From Time Zero to Time 't' (AUC[0-t]) Following Intravenous (IV) and Subcutaneous (SC) JNJ-61178104 Administration | Up to Day 113
Area Under the Serum Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) Following Intravenous (IV) and Subcutaneous (SC) JNJ-61178104 Administration | Up to Day 113
Serum Half-Life (t1/2) Following Intravenous (IV) and Subcutaneous (SC) JNJ-61178104 Administration | Up to Day 113
Time to Reach Maximum Observed Serum Concentration (Tmax) Following Subcutaneous (SC) JNJ-61178104 Administration | Up to Day 113
Systemic Clearance (CL) Following Intravenous (IV) JNJ-61178104 Administration | Up to Day 113
Apparent Clearance (CL/F) Following Subcutaneous (SC) JNJ-61178104 Administration | Up to Day 113
Volume of Distribution (Vz) Following Intravenous (IV) JNJ-61178104 Administration | Up to Day 113
Apparent Volume of Distribution (Vz/F) Following Subcutaneous (SC) JNJ-61178104 Administration | Up to Day 113
Absolute Bioavailability (F[abs]) Following Subcutaneous (SC) JNJ-61178104 Administration | Up to Day 113
  The F is the percentage of the subcutaneously administered dose that is systemically available relative to an intravenous (IV) administration. It is calculated as (AUC [0-infinity] for 1 mg/kg SC JNJ-61178104)/(AUC [0-infinity] for 1 mg/kg IV JNJ-61178104 )*100, where the AUC (0-infinity) is area under the concentration-time curve from time zero to extrapolated infinite time.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium